CLINICAL TRIAL: NCT00309920
Title: Adjuvant Therapy of Breast Cancer: Impact of Erythropoiesis Stimulating Factors on Event Free Survival High Risk Breast Cancer Treatment
Brief Title: Combination Chemotherapy With or Without Darbepoetin Alfa in Treating Women With Stage III Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000458037; WGSG-ARA-PLUS; AVENTIS-WGSG-ARA-PLUS; SANOFI-WGSF-ARA-PLUS; EU-205108
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2006-04

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Darbepoetin alfa; Cyclophosphamide; Docetaxel; Doxorubicin; Epirubicin; Fluorouracil

INTERVENTIONS:
Biological: darbepoetin alfa
Drug: cyclophosphamide
Drug: docetaxel
Drug: doxorubicin hydrochloride
Drug: epirubicin hydrochloride
Drug: fluorouracil

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Colony-stimulating factors, such as darbepoetin alfa, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy. Giving combination chemotherapy together with darbepoetin alfa after surgery may kill any tumor cells that remain after surgery. It is not yet known whether combination chemotherapy and darbepoetin alfa are more effective than combination chemotherapy alone in treating stage III breast cancer.

PURPOSE: This randomized clinical trial is studying how well giving combination chemotherapy together with darbepoetin alfa works compared to combination chemotherapy alone in treating women with stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the disease-free survival rate in women with stage III breast cancer treated with adjuvant chemotherapy with vs without darbepoetin alfa.

Secondary

* Compare local recurrence and overall survival in patients receiving these regimens.
* Compare toxicity of these regimens in these patients.
* Compare quality of life and fatigue frequency in patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according the chemotherapy regimen (CEF vs TAC). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive 1 of the following regimens:

  * Regimen CEF: Patients receive cyclophosphamide IV, epirubicin hydrochloride IV, and fluorouracil IV on day 1.
  * Regimen TAC: Patients receive docetaxel IV, doxorubicin hydrochloride IV, and cyclophosphamide IV on day 1.

Treatment repeats every 3 weeks for 6 courses in the absence of disease progression and unacceptable toxicity.

* Arm II: Patients receive 1 of the following regimens:

  * Regimen CEF: Patients receive regimen CEF as in arm I. Patients receive darbepoetin alfa if hemoglobin falls to ≤ 13.0 g/dL. Darbepoetin alfa is discontinued when hemoglobin rises to > 14.0 g/dL.
  * Regimen TAC: Patients receive TAC as in arm I and darbepoetin alfa as in arm II, regimen CEF.

Quality of life is assessed at baseline, before each chemotherapy course, at the completion of study therapy, and at 6 and 12 months.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 1,234 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Stage III disease (pT1, N2-3, M0)
  * No metastatic disease by thoracic x-ray, full-body bone scan, and liver sonography
* No inflammatory disease or Paget's disease
* Disease completely resected (R0) and ≥ 10 axillary lymph nodes removed

  * Underwent surgery approximately 42 days ago
  * At least 9 positive lymph nodes
  * No prior sequential mastectomy
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* ECOG performance status 0-1
* WBC ≥ 3,500/mm^3
* Creatinine ≤ 1.4 mg/dL
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 2.0 mg/dL
* No pre-existing symptomatic peripheral neuropathy
* Not pregnant or nursing
* No hypersensitivity to darbepoetin alfa, epoetin alfa, or any of their components
* No other malignancy except curatively treated basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No participation in another clinical study
* No prior therapies that would preclude study participation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1234 (Estimated)
Dates: Start 2004-01

PRIMARY OUTCOMES:
Disease-free survival at 6 months to 5 years after treatment

SECONDARY OUTCOMES:
Overall survival at 6 months to 5 years after treatment
Toxicity by NCI toxicity criteria at every course and periodically thereafter
Anemia and cognitive function by Functional Assessment of Cancer Therapy-Cognitive (FACT-Cog) at every course
Local relapses at 6 months to 5 years after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Nitz, PhD, Study Chair — Heinrich-Heine University, Duesseldorf
Locations (47):
- Germany (47):
  - Kreiskrankenhaus Aurich, Aurich
  - Maria-Hilf-Krankenhaus, Bergheim
  - Evangelisches Krankenhaus - Bergisch Gladbach, Bergisch
  - Johanniter-Krankenhaus Bonn, Bonn
  - Onkologische Gemeinschaftspraxis, Bonn
  - Praxis fuer Haematologie - Onkologie, Bonn-Duisdorf
  - St. Rochus Hospital, Castrop-Rauxel
  - Praxis Fuer Haematologie Internistische Onkologie, Cologne
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - St. Elisabeth-Krankenhaus - Koeln, Cologne
  - Klinikum Deggendorf, Deggendorf
  - Onkologische Schwerpunktpraxis, Duisburg
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Alfried Krupp Krankenhaus, Essen
  - Universitaetsklinikum Essen, Essen
  - II Medizinische Klinik - Klinikum Fuerth, Fürth
  - Evangelische Kliniken Gelsenkirchen GmbH, Gelsenkirchen
  - Wilhelm-Anton-Hospital gGmbH, Goch, Goch
  - Maria-Josef-Hospital Greven GmbH, Greven
  - Allgemeines Krankenhaus Hagen, Hagen
  - Evangelisches Krankenhaus Hagen-Haspe GmbH, Hagen
  - Henriettenstiftung Krankenhaus, Hanover
  - Praxisgemeinschaft fuer Gynaekologische Onkologie, Hildesheim
  - Universitaetsklinikum des Saarlandes, Homburg
  - Klinikum Kaufbeuren Ostallgaeu, Kaufbeuren
  - Katholisches Klinikum Koblenz Marienhof, Koblenz
  - Frankenwald Klinik, Kronach
  - Internistische Onkologische Praxis - Kronach, Kronach
  - Knappschaft Krankenhaus, Langendreer
  - St. Marien Hospital - Luenen, Lünen
  - St. Vincenz und Elisabeth Hospital, Mainz
  - Klinikum Memmingen, Memmingen
  - Klinikum Minden, Minden
  - Krankenhaus Bethanien, Moers
  - Marienhaus Klinikum St. Elisabeth Neuwied, Neuwied
  - Evangelisches Krankenhaus Oberhausen, Oberhausen
  - Internistische Gemeinschaftspraxis - Offenbach, Offenbach
  - Praxis fuer Haematologie und Onkoligie, Rheine
  - Klinikum Suedstadt Rostock, Rostock
  - Marienkrankenhaus Schwerte gem. GmbH, Schwerte
  - Staedtisches Klinikum Solingen, Solingen
  - Praxis Fuer Internistische Haematologie / Onkologie, Troisdorf
  - Katherinen-Hospital gGmbH, Unna
  - Marien-Hospital Wesel gGmbH, Wesel
  - Marien-Hospital Witten, Witten
  - Bethesda Krankenhaus Wuppertal gGmbH, Wuppertal
  - Haematologie / Onkologische Schwerpunktpraxis, Wuppertal